CLINICAL TRIAL: NCT02345148
Title: An Open-Label, Single-Dose Study to Assess the Pharmacokinetics, Safety, and Tolerability of Intranasally Administered Esketamine in Elderly (>= 75 Years of Age) and Healthy Younger Adult Subjects (18 to 55 Years of Age, Inclusive)
Brief Title: Pharmacokinetic, Safety, and Tolerability Study of Intranasally Administered Esketamine in Elderly and and Healthy Younger Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR106172; ESKETINTRD1012 (Other: Janssen Research & Development, LLC); 2014-003690-42 (EudraCT Number)
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Healthy
Keywords: Healthy; Esketamine; JNJ-54135419
MeSH Terms: interventions — Esketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Elder participants will receive esketamine hydrochloride solution (containing 14 milligram (mg) of esketamine base per 100 microliter [mcl] of intranasal spray) by intranasal route using nasal spray pump at 0, 5 and 10 minutes on Day 1.
  Interventions: Drug: Esketamine
- Cohort 2 (Experimental): Younger adults will receive esketamine hydrochloride solution (containing 14 milligram (mg) of esketamine base per 100 microliter [mcl] of intranasal spray) by intranasal route using nasal spray pump at 0, 5 and 10 minutes on Day 1.
  Interventions: Drug: Esketamine

INTERVENTIONS:
Drug: Esketamine — Esketamine 84 mg will be self-administered by participants as intranasal spray at 0, 5 and 10 minutes on Day 1.
  Other Names: Esketamine hydrochloride; JNJ-54135419

SUMMARY:
The purpose of this study is to compare the pharmacokinetics, safety, and tolerability of intranasally administered esketamine in elderly participants (greater than equal to [>=] 75 years of age) and younger healthy adult participants (18 to 55 years of age, inclusive).

DETAILED DESCRIPTION:
This is a single-center, 2-cohort, single-dose, open-label study. The duration of study will be approximately 42 days per participant. The study consists of 3 parts: Screening (that is, 28 days before study commences on Day 1) and open-label Treatment (Day 1) and Follow-up (up to Day 13). Esketamine will be administered by intranasal route (delivery of medications through the nasal mucosa) on Day 1. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* For Cohort 1, be a man or woman, >= 75 years of age who are either healthy or who present with stable, well-controlled, chronic conditions which frequently occur in the elderly, such as: hyperlipidemia; controlled hypertension; impaired fasting glucose, impaired glucose tolerance or type 2 diabetes mellitus controlled with diet, and/or metformin monotherapy, dipeptidyl peptidase-4 (DPP-4) inhibitor monotherapy or a combination of metformin and DPP-4 inhibitor, who have glycated hemoglobin (HbA1c) levels less than 8 percent; degenerative joint disorders and osteoporosis; kidney function decline appropriate for age. Inclusion of participants with other chronic, well-controlled and stable conditions to Cohort 1 should be reviewed and agreed between the Investigator and the Sponsor
* For Cohort 2, be a man or woman, 18 to 55 years of age, inclusive
* For women of childbearing potential in Cohort 2, must have a negative serum beta-human chorionic gonadotropin (hCG) pregnancy test at screening; and a negative urine pregnancy test on Day -1
* If a man, must agree to use an adequate contraception method as deemed appropriate by the investigator and to not donate sperm during the study and for 3 months after receiving the study drug
* Body mass index (BMI) (weight [kg]/height^2 [m]^2) between 18 and 32 kg/m^2 (inclusive), and body weight not less than 50 kg

Exclusion Criteria:

* Diagnosed with a current or previous psychiatric disorder including but not limited to psychotic, bipolar, major depressive, or anxiety disorder
* Clinically significant medical illness
* Severe renal impairment
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening or at admission to the study center (Day -1) as deemed appropriate by the investigator
* History of drug or alcohol abuse disorder within the past 1 year, or a reason to believe a participant has such a history

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | up to 24 hours after study drug administration
  The Cmax is the maximum plasma concentration.
Time to reach maximum concentration (tmax) | up to 24 hours after study drug administration
  The Tmax is time to reach the maximum plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to 12 Hours (AUC [0-12]) | up to 24 hours after study drug administration
  The AUC (0-12) is the area under the plasma concentration-time curve from time 0 to 12 hours post-dose.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last (AUC [0-last]) | up to 24 hours after study drug administration
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time, calculated as the sum of AUC(last) and C(last)/lambda(z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; and C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | up to 24 hours after study drug administration
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; and C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Elimination half-life period (t1/2) associated with the terminal slope (Lambda z) | up to 24 hours after study drug administration
  Elimination half-life associated with the terminal slope (lambda[z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/lambda(z).
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | 42 days
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium

REFERENCES:
- [Derived] Perez-Ruixo C, Rossenu S, Zannikos P, Nandy P, Singh J, Drevets WC, Perez-Ruixo JJ. Population Pharmacokinetics of Esketamine Nasal Spray and its Metabolite Noresketamine in Healthy Subjects and Patients with Treatment-Resistant Depression. Clin Pharmacokinet. 2021 Apr;60(4):501-516. doi: 10.1007/s40262-020-00953-4. Epub 2020 Oct 31. PMID 33128208